CLINICAL TRIAL: NCT02211742
Title: Short-term Effects of Dapagliflozin on Fasting and Postprandial Glucose Homeostasis in Male Type 1 Diabetes Patients.
Brief Title: Dapagliflozin in Type 1 Diabetes
Acronym: DapaT1DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Collaborators: Medical University of Graz (Other); University of Bern (Other)
Responsible Party: Principal Investigator, Markus Laimer, PD MD, Medical University Innsbruck
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CUI_001
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Fasting Glucose; Glucose Excursion; Glycemic Control
Keywords: dapagliflozin; fasting glucose; postprandial glucose excursion; euglycemic hyperinsulinemic clamp; euglycemic oral glucose tolerance test
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dapagliflozin (Active Comparator): 10mg dapagliflozin per 24h for 3 days per cross-over phase (equals 2 x 30mg)
  Interventions: Drug: Dapagliflozin
- placebo sugar pills (Placebo Comparator): placebo tablet, 1 per 24h for 3 days in total per cross-over phase (equals 2 x 3 tablets)
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — euglycemic hyperinsulinemic clamp tests and euglycemic oral glucose tolerance clamp tests after the short-term (i.e.: 3 days, equals 10mg / 24h) intake of dapagliflozin

SUMMARY:
Dapagliflozin is a highly selective, reversible and potent inhibitor of the sodium-glucose-linked Transporter 2 (SGLT2), which was successfully investigated for its use as a treatment option in type 2 diabetes mellitus. The effect of dapagliflozin is an increased glucosuria, and it was shown that mean blood glucose concentrations and postprandial glucose excursion in special were significantly reduced in type 2 diabetic patients. Due to its mechanism-of action it seems likely that also type 1 diabetic patients will benefit from dapagliflozin. The present study is focused on the effects of dapagliflozin on fasting glucose homeostasis and postprandial glucose excursion in male type 1diabetic patients. Participants will subsequently receive 10 milligrams of dapagliflozin and placebo for 3 days (equals 2 x 30mg per cross-over period) in a double-blind, randomised, cross-over design. The effects will be measured via euglycemic hyperinsulinemic clamp studies (fasting glucose homeostasis) and euglycemic oral glucose tolerance clamp tests (postprandial glucose excursions).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (duration of disease at least 5 years)
* C-peptide concentration < 0.2µg/l
* male sex
* aged 18 to 60 years
* Body Mass Index 20 - 25 kg/m2
* no measurable, clinically relevant ketonuria

Exclusion Criteria:

* insufficient venous status on both forearms
* renal and/or hepatic insufficiency (including microalbuminuria and/or albumin/creatinin-ratio)
* history of cancer
* intake of medication and/or substances capable to influence insulin sensitivity within the last 3 months prior to study inclusion
* alcohol- and/or drug abuse, nicotine consumption > 5 cigarettes / 24h
* brittle-diabetes
* history of severe hypoglycemia, defined as the need for foreign assistance independent of actual blood glucose concentration measured
* history or evidence of any other clinically significant disorder, condition or disease other than those outlined above that, in the opinion of the investigator may compromise the ability of the participant to give written informed consent, would pose a risk to subject safety, or interfere with the study evaluation, procedures or completion.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
fasting glucose homeostasis | study visit, immediatly
  During hyperinsulinemic, euglycemic clamp studies, fasting glucose homeostasis will be determined for both, dapagliflozin and placebo.
postprandial glucose homeostasis | study visit, immediatly
  During euglycemic oral glucose tolerance clamp tests, postprandial glucose excursion will be determined and compared between dapagliflozin and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Laimer, PD MD, Principal Investigator — Medical University Innsbruck, Department of Internal Medicine I
Locations (1):
- Medical University Innsbruck, Department of Internal Medicine I, Innsbruck, Tyrol, Austria

REFERENCES:
- [Background] DeFronzo RA, Hompesch M, Kasichayanula S, Liu X, Hong Y, Pfister M, Morrow LA, Leslie BR, Boulton DW, Ching A, LaCreta FP, Griffen SC. Characterization of renal glucose reabsorption in response to dapagliflozin in healthy subjects and subjects with type 2 diabetes. Diabetes Care. 2013 Oct;36(10):3169-76. doi: 10.2337/dc13-0387. Epub 2013 Jun 4. PMID 23735727
- [Background] Abdul-Ghani MA, DeFronzo RA. Dapagliflozin for the treatment of type 2 diabetes. Expert Opin Pharmacother. 2013 Aug;14(12):1695-703. doi: 10.1517/14656566.2013.812632. Epub 2013 Jun 26. PMID 23800130
- [Background] Mather A, Pollock C. Glucose handling by the kidney. Kidney Int Suppl. 2011 Mar;(120):S1-6. doi: 10.1038/ki.2010.509. PMID 21358696
- [Background] Plosker GL. Dapagliflozin: a review of its use in type 2 diabetes mellitus. Drugs. 2012 Dec 3;72(17):2289-312. doi: 10.2165/11209910-000000000-00000. PMID 23170914